CLINICAL TRIAL: NCT06895343
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single Ascending Doses of ABBV-701 in Healthy Adult Western and Asian Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single Ascending Subcutaneous or Intravenous Doses of ABBV-701 in Healthy Adult Western and Asian Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M25-491
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-701

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part 1: Group 1 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose A or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 1: Group 2 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose B or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 1: Group 3 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose C or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 1: Group 4 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose D or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 1: Group 5 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose E or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 2: Group 6 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose E or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 2: Group 7 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose E or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 3: Group 8 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose C or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 3: Group 9 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose E or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 3: Group 10 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose F or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 4: Group 11 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose F or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo
- Part 4: Group 12 ABBV-701 or Placebo (Experimental): Participants will receive a single dose of either ABBV-701 Dose F or placebo.
  Interventions: Drug: ABBV-701; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-701 — Subcutaneous
  Arms: Part 1: Group 1 ABBV-701 or Placebo; Part 1: Group 2 ABBV-701 or Placebo; Part 1: Group 3 ABBV-701 or Placebo; Part 1: Group 4 ABBV-701 or Placebo; Part 1: Group 5 ABBV-701 or Placebo; Part 2: Group 6 ABBV-701 or Placebo; Part 2: Group 7 ABBV-701 or Placebo
Drug: Placebo — Subcutaneous
  Arms: Part 1: Group 1 ABBV-701 or Placebo; Part 1: Group 2 ABBV-701 or Placebo; Part 1: Group 3 ABBV-701 or Placebo; Part 1: Group 4 ABBV-701 or Placebo; Part 1: Group 5 ABBV-701 or Placebo; Part 2: Group 6 ABBV-701 or Placebo; Part 2: Group 7 ABBV-701 or Placebo
Drug: ABBV-701 — IV Infusion
  Arms: Part 3: Group 10 ABBV-701 or Placebo; Part 3: Group 8 ABBV-701 or Placebo; Part 3: Group 9 ABBV-701 or Placebo; Part 4: Group 11 ABBV-701 or Placebo; Part 4: Group 12 ABBV-701 or Placebo
Drug: Placebo — IV infusion
  Arms: Part 3: Group 10 ABBV-701 or Placebo; Part 3: Group 8 ABBV-701 or Placebo; Part 3: Group 9 ABBV-701 or Placebo; Part 4: Group 11 ABBV-701 or Placebo; Part 4: Group 12 ABBV-701 or Placebo

SUMMARY:
The main objective of this study is to assess the safety, tolerability, pharmacokinetics, and immunogenicity of single ascending doses of ABBV-701 in healthy adult western and Asian participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight is ≥ 35 kg and BMI is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenth's decimal.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG
* Part 2 and Part 4 only:

For Japanese Participants:

--Participant must be first or second-generation Japanese parentage (both parents of Japanese descent), residing outside of Japan. Participants must be in general good health and maintain a typical Japanese lifestyle, including consuming a typical Japanese diet.

Han Chinese Participants:

--Participant must be first or second-generation Han Chinese of full Chinese parentage (both parents of Han Chinese descent), residing outside of China. Participants must be in general good health and maintain a typical Chinese lifestyle, including consuming a typical Chinese diet.

Exclusion Criteria:

* History of any clinically significant cardiovascular, respiratory (except mild asthma as a child), renal, endocrine, hepatic, gastrointestinal, hematologic, or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 47 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Plasma Concentration (Cmax) of ABBV-701 | Up to approximately 47 weeks
  Cmax of ABBV-701
Time to Cmax (Tmax) of ABBV-701 | Up to approximately 47 weeks
  Tmax of ABBV-701
Apparent terminal phase elimination rate constant (β) of ABBV-701 | Up to approximately 47 weeks
  (β) of ABBV-701
Terminal Phase Elimination Half-Life (t1/2) of ABBV-701 | Up to approximately 47 weeks
  (t1/2) of ABBV-701
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-701 | Up to approximately 47 weeks
  AUCt of ABBV-701
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-701 | Up to approximately 47 weeks
  AUCinf of ABBV-701

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - CenExel ACT- Anaheim Clinical Trials /ID# 278431, Anaheim, California
  - Acpru /Id# 273354, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-491